CLINICAL TRIAL: NCT01892176
Title: Effects of High-dose Coenzyme Q10 on Biomarkers of Oxidative Damage and Clinical Outcome in Parkinson Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Associate Professor, National University Hospital, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB/2010/00223
Record Dates: First submitted 2013-06-30; First posted 2013-07-04 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Parkinson Disease
Keywords: coenzyme Q10, Parkinson disease, oxidative damage
MeSH Terms: conditions — Parkinson Disease | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coenzyme Q10 (Experimental): 400mg/day, 800mg/day, 1200/day and 2400mg/day
  Interventions: Dietary Supplement: coenzyme q10

INTERVENTIONS:
Dietary Supplement: coenzyme q10 — 400mg/day, 800mg/day, 1200/day and 2400mg/day

SUMMARY:
The investigators hypothesise that measuring biomarkers of oxidative damage could better inform investigators on the potential merits (and pitfalls) of CoQ10 supplementation in PD subjects.

DETAILED DESCRIPTION:
Subjects with idiopathic PD will be recruited to a 10-week dose escalation study. Each dosage (400mg/day, 800mg/day, 1200/day and 2400mg/day) will be consumed daily for two weeks. Information on safety and fasting blood/urine samples will be collected. Primary endpoint is plasma F2-isoprostanes (adjusted for arachidonate) while secondary endpoint is the change in the total Unified Parkinson Disease Rating Scale (UPDRS) before and after treatment. Serum phospholipase A2 activities, plasma all trans-retinol, plasma total tocopherol (sum of α-, δ- and γ-tocopherol) and serum uric acid will be measured.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson disease
* age >21 years
* able to provide written informed consent

Exclusion Criteria:

* diabetes mellitus, stroke, cardiac and renal diseases and cigarette smoking
* major psychiatric disorder or drug and/or alcohol abuse/dependence
* regular use of antioxidants, dietary supplements, traditional Chinese remedies, non-steroidal anti-inflammatory drugs or immunosuppressive drugs

Min Age: 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers of oxidative damage | 10 weeks

SECONDARY OUTCOMES:
Total Unified Parkinson's Disease Rating Scale (UPDRS) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Seet, MBBS, Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore, Singapore